CLINICAL TRIAL: NCT06387563
Title: Effects of Abdominal Muscle Activation Training, Using Pressure Biofeedback in Comparison With Surface Electromyography
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Foundation University Islamabad (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FUI/CTR/2024/4
Record Dates: First submitted 2024-04-23; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Randomized control trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Abdominal activation using pressure biofeedback (Experimental): Group A PBF assisted abdominal muscle activation training (30 min, 3x /week /4 weeks) Progressive Muscle Relaxation for 5 min Pressure biofeedback assisted abdominal muscle activation training. Frequency: 25 min; 10 sec hold, 15 sec relax, 10 reps Progression criteria in training: Maintaining 3 - 5 mmHg pressure on PBF dial while performing abdominal muscle activation.
  Exercises for Group For biofeedback assisted abdominal muscle activation training these exercises will be performed:
  1. Supine abdominal muscle activation (45° Hip knee flexion)
  2. Both hip and knee 90° flexion
  3. One side hip and knee 90° flexion with other fully extended
  4. One side hip and knee 90° flexion with other fully extended + heel 12 cm raised
  5. Both legs fully extended with heel 12 cm raised
  6. Partial curl ups
  7. Prone lying abdominal muscle activation
  8. Prone leg raises
  9. Prone upper back extension simple
  10. Prone reciprocal UE/LE exercises
  Interventions: Procedure: Abdominal activation using pressure biofeedback
- Group B: Abdominal activation using SEMG biofeedback (Experimental): GROUP B:
  SEMG-BF assisted abdominal muscle activation training (30 min, 3x/ week/ 4 weeks) Progressive Muscle Relaxation for 5 min Surface EMG-BF assisted abdominal muscle activation training. Frequency: 25 min; 10 sec hold, 15 sec relax, 10 reps Maintaining minimal volumetric contraction of abdominal muscle activation (as per person) on SEMG device with abdominal muscle activation for set frequency
  Exercises for Group B For biofeedback assisted abdominal muscle activation training these exercises will be performed:
  1. Supine abdominal muscle activation (45° Hip knee flexion)
  2. Both hip and knee 90° flexion
  3. One side hip and knee 90° flexion with other fully extended
  4. One side hip and knee 90° flexion with other fully extended + heel 12 cm raised
  5. Both legs fully extended with heel 12 cm raised
  6. Partial curl ups
  7. Prone lying abdominal muscle activation
  8. Prone leg raises
  9. Prone upper back extension simple
  10. Prone reciprocal UE/LE exercises
  Interventions: Procedure: Abdominal activation using SEMG biofeedback

INTERVENTIONS:
Procedure: Abdominal activation using pressure biofeedback — PBF assisted abdominal muscle activation training (30 min, 3x /week /4 weeks) Progressive Muscle Relaxation for 5 min Pressure biofeedback assisted abdominal muscle activation training. Frequency: 25 min; 10 sec hold, 15 sec relax, 10 reps Progression criteria in training: Maintaining 3 - 5 mmHg pressure on PBF dial while performing abdominal muscle activation.
  Exercises for Group For biofeedback assisted abdominal muscle activation training these exercises will be performed:
  1. Supine abdominal muscle activation (45° Hip knee flexion)
  2. Both hip and knee 90° flexion
  3. One side hip and knee 90° flexion with other fully extended
  4. One side hip and knee 90° flexion with other fully extended + heel 12 cm raised
  5. Both legs fully extended with heel 12 cm raised
  6. Partial curl ups
  7. Prone lying abdominal muscle activation
  8. Prone leg raises
  9. Prone upper back extension simple
  10. Prone reciprocal UE/LE exercises
  Arms: Group A: Abdominal activation using pressure biofeedback
Procedure: Abdominal activation using SEMG biofeedback — SEMG-BF assisted abdominal muscle activation training (30 min, 3x/ week/ 4 weeks) Progressive Muscle Relaxation for 5 min Surface EMG-BF assisted abdominal muscle activation training. Frequency: 25 min; 10 sec hold, 15 sec relax, 10 reps Maintaining minimal volumetric contraction of abdominal muscle activation (as per person) on SEMG device with abdominal muscle activation for set frequency
  Exercises for Group B For biofeedback assisted abdominal muscle activation training these exercises will be performed:
  1. Supine abdominal muscle activation (45° Hip knee flexion)
  2. Both hip and knee 90° flexion
  3. One side hip and knee 90° flexion with other fully extended
  4. One side hip and knee 90° flexion with other fully extended + heel 12 cm raised
  5. Both legs fully extended with heel 12 cm raised
  6. Partial curl ups
  7. Prone lying abdominal muscle activation
  8. Prone leg raises
  9. Prone upper back extension simple
  10. Prone reciprocal UE/LE exercises
  Arms: Group B: Abdominal activation using SEMG biofeedback

SUMMARY:
This study is a randomized control trial and the purpose of this study to determine the effects of abdominal muscle activation training on non-specific low back pain; using pressure biofeedback in comparison with surface electromyography biofeedback: a randomized control trial.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effects of abdominal muscle activation training, using pressure biofeedback in comparison with surface electromyography biofeedback, in management of non-specific low back pain: a randomized control trial.

Pain and disability are the primary outcomes which will be determined using:

1. Numeric pain rating scale (NPRS)
2. Oswestry disability index (ODI) Data will be taken before and after the intervention protocol for each participant.

Data collection procedure: Participants of interest would be approached and explained about the research. Informed written consent will be taken. Pre and post intervention scores will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age (adults 19 - 44 years)
* Non-specific LBP with NPRS > 3
* Negative SLR test in prone and supine
* Painless extremity movement and activity
* Manual muscle testing of abdominal muscles between grade 2 - 4
* Sedentary individuals (no exercise plan followed in last 3 months)

Exclusion Criteria:

* History of any spinal surgery
* Degenerative disc disorder, facet joint syndrome, spinal stenosis, myelopathy, lumbar syringomyelia
* Sensory disturbances due to neurological causes, lumbar radiculopathy, fibromyalgia, myofascial pain syndrome
* Sacroiliac joint dysfunction
* Pregnancy
* Medical conditions; Hypertension, Diabetes mellites
* Work disability greater than 6 months
* Not able to attend regular therapy appointments

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-06 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | 4 weeks
  The NPRS will be used to quantify LBP, and it exhibits good validity ranging from 0.79 to 0.95, as well as reliability ranging from 0.67 to 0.96(23). The scoring for NPRS involves a scale from 0 to 10, where 0 indicates no pain. The interpretation of scores is as follows: 0 to 3 for mild pain, 4 to 6 for moderate pain, and 7 to 10 for severe pain.
Level of Disability | 4 weeks
  For measuring disability, Oswestry Disability Index will be utilized

CONTACTS AND LOCATIONS:
Locations (1):
- Foundation University College of Physical Therapy, Rawalpindi, Punjab Province, Pakistan